CLINICAL TRIAL: NCT03517072
Title: Determinants of the Long-Term Success of Bariatric Surgery "- Multicenter Regional Observational Study: Regional Multicentre Prospective Study
Brief Title: Determinants of the Long-Term Success of Bariatric Surgery
Acronym: PRECOS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2016_24; 2016-A02058-43 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-04-24; First posted 2018-05-07 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Morbid Obesity; Bariatric Surgery Candidate
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The management of obesity is based on a multidisciplinary approach and justifies the use of surgery in patients with the most severe forms. Surgery for obesity or bariatric surgery generally allows rapid and significant weight loss however it is associated with significant risks, and its long-term results remain heterogeneous and unpredictable. Long-term data will clarify the role of different types of bariatric surgery in surgical strategy, improve patient information and identify predictors of failure in order to provide personalised and tailored surgery for each candidate .

DETAILED DESCRIPTION:
Currently, there is insufficient data to determine the persistence over time of the positive results of bariatric surgery on weight loss. Moreover, there is no consensus or criteria for choosing one surgical weight loss procedure over another. The best choice for one patient may not be the most appropriate for another.

The results of this project will allow to better select obese patients likely to benefit from bariatric surgery, and to further personalise the management of severe obesity.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received bariatric surgery 5 years ago.

Exclusion Criteria:

* Refusal to participate in the study,
* Unable to receive informed information,
* Unable to participate in the study

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The project relies on the network of Specialised Centres for the Management of Severe Obesity (Lille, Arras, Boulogne, Valenciennes).
  Patients with severe obesity who underwent bariatric surgery 5 years ago will be included in each of the centre, during the usual multidisciplinary care visit.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-07-31 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Success rate in terms of weight loss | at 5 years after bariatric surgery
  Rate of patients who lost at least 20 of their initial body weight

SECONDARY OUTCOMES:
Success rate in terms of weight loss according to type of bariatric surgery | at 1 year after bariatric surgery
  Rate of patients who lost at least 20 of their initial body weight at 1 year according to type of bariatric surgery (Gastric by-pass in Y or Omega, sleeve gastrectomy, and gastric band)
Success rate in terms of weight loss according to type of bariatric surgery | at 5 years after bariatric surgery
  Rate of patients who lost at least 20 of their initial body weight at 5 years according to type of bariatric surgery (Gastric by-pass in Y or Omega, sleeve gastrectomy, and gastric band)
Rate of re- interventions related to bariatric surgery | 5 years
  Evaluation of re-interventions following bariatric surgery
Lost rate seen | at 5 years after bariatric surgery
  Evaluation of lost to follow-up

CONTACTS AND LOCATIONS:
Overall Officials: François PATTOU, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (4):
- France (4):
  - CH ARRAS, Arras
  - Ch Boulogne-Sur-Mer, Boulogne-sur-Mer
  - Hôpital Claude Huriez, CHU, Lille
  - Ch de Valenciennes, Valenciennes